CLINICAL TRIAL: NCT04177420
Title: Investigation for Health Efficacy of Infrared-C Radiation on Diabetes Patients in Senior's Activity Center
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanhua University (Other)
Collaborators: Buddhist Dalin Tzu Chi General Hospital (Unknown); Solano Semiconductor Technology., LTD. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: B10701016
Record Dates: First submitted 2019-06-08; First posted 2019-11-26 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Types 2 Diabetes Mellitus; Glycation; AGEs; hemoglobin A1c, HbA1c; Fasting blood sugar, GLU-AC; Insulin; Procollagen-I N-telopeptide, PINP; C-telopeptide of type I collagen, CTx; osteocalcin; Pittsburgh sleep quality index, PSQI; numeric rating scale-knee, NRS-knee; Geriatric depression Scale-15, GDS-15; Total Antioxidant Capacity, TAC; Infrared-C; Hyperglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance; Xanthomatosis, Cerebrotendinous; Hyperglycemia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experiment Group (Experimental): lay on the FIR-C mattress with cover the FIR-C abdominal pad on abdominal part and Knee part during the sleeping time. The controller will switch on and switch off rotated in each hour for whole night.
  Interventions: Device: FIR-C mattress; Device: FIR-C abdominal pad
- Control Group (Placebo Comparator): lay on the FIR-C mattress with cover the FIR-C abdominal pad on abdominal part and Knee part during the sleeping time. The controller will switch on and switch off rotated in each hour for whole night. the FIR-C mattress and the FIR-C abdominal pad is malfunction and it can not produce the FIR-C.
  Interventions: Device: fake FIR-C mattress; Device: fake FIR-C abdominal pad

INTERVENTIONS:
Device: FIR-C mattress — infrared-C irradiation by hot mattress with a powered heating compress
  Arms: Experiment Group
Device: FIR-C abdominal pad — infrared-C irradiation by hot abdominal pad with a powered heating compress
  Arms: Experiment Group
Device: fake FIR-C mattress — normal mattress with fake controller, custom make for placebo group
  Arms: Control Group
Device: fake FIR-C abdominal pad — normal abdominal pad with fake controller, custom make for placebo group
  Arms: Control Group

SUMMARY:
Hyperglycemia caused by diabetes will bring us the long-term damage，it causes glycation. The combination of sugar molecules and protein molecules will transform to advanced glycation end products (AGEs) and produce a lot of free radicals to caused inflammatory reactions, forming various comorbidities, affecting the function of different organs, especially the eyes, kidneys, nervous system, heart, blood vessels and damage to bone structure and bone Quality, which leads to bone loss. Therefore, the development of alternative therapies is important for the treatment of diabetes. We assume the 4 months experiment can normalize subjects HbA1c.

DETAILED DESCRIPTION:
In the past research from our team, it was found that far infrared ray (FIR) helps to reduce oxidative stress in the body and is expected to contribute to the treatment of diabetes. Therefore, the team hopes to effectively reduce glycated hemoglobin (HbA1c), fasting blood glucose (GLU-AC), insulin (insulin), reduce the body's oxidative stress index, increase Total Antioxidant Capacity (TAC) inhibit the inflammatory response and reduce complications through 4 months of IR-C intervention. Which expected to reduce the index of the nitrogen-type first collagen element (Procollagen-I N -telopeptide, PINP) and C-telopeptide of type I collagen (CTx) bone loss index, enhance Osteocalcin's index of bone growth indicators. Along with the Pittsburgh sleep quality index (PSQI), numeric rating scale-knee (NRS-knee) and Geriatric depression Scale-15 (GDS-15) to reduce the number of times the elderly take medication and improve their health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c higher than 6.8% or fasting blood sugar higher than 126mg/dL;
* Conscious, mental and cognitively normal;
* no obstacles in action;
* can read, write and communicate with mandarin, taiwanese and hakka.

Exclusion Criteria:

* Inflammatory skin wounds on the neck, back, lower back or lower leg;
* obstacles in communication;
* People with disabilities, epilepsy, and other unacceptable warming treatments;
* When the subject finds that he or she is unwell during the procedure, the experiment is terminated and take care by the medical staff.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-15 (Estimated)

PRIMARY OUTCOMES:
Hemoglobin A1c, HbA1c | Baseline to 4 months
  The hemoglobin A1c can show us our average level of blood sugar over the past 2 to 3 months. Below 6% is normal, over 6% is abnormal.
Fasting Blood Sugar, GLU-AC | Baseline to 4 months
  A blood sample will be taken after an overnight fast which to estimate blood sugar levels. Below 100mg/dL is normal, 100 to 125mg/dL is prediabetes, 125mg/dL above is consider diabetes.
Insulin | Baseline to 4 months
  Is a hormone that is produced and stored in the beta cells of the pancreas. this test can measures the amount of insulin in the blood which to analyze the insulin resistance of the body.
Superoxide, O2- | Baseline to 4 months
  superoxide is one type of the free radical. The assay of superoxide can show us the ability to inhibit free radical contained in blood. The highest value of it means the highest injured did. The data of the post-test should be lower than the data of the pre-test.
Osteocalcin | Baseline to 4 months
  Is a noncollagenous protein hormone found in bone and dentin, it implicated in bone mineralization and calcium ion homeostasis. The normal range for female: 12-23ng/dL; the normal range for male: 17-26ng/dL.
Procollagen-I N-telopeptide, PINP | Baseline to 4 months
  This market is a specific indicator of type I collagen deposition therefore can set as an indicator of bone formation velocity. The reference's range for PINP: 16.27 - 73.87 ng/mL.
C-telopeptide of type I collagen，CTx | Baseline to 4 months
  It is the carbon-terminal fragment of the first type of collagen in the bone, which is the final product of bone decomposition and can be used as an indicator of bone loss. The reference's range for female: 0.104-1.008ng/mL; for male: 0.000-0.854ng/mL
Total Antioxidant Capacity, TAC | Baseline to 4 months
  to assess the antioxidant status of blood to evaluate the antioxidant response against the free radicals produced in the blood. The reference's range for male: >=0.65mmol/L; female: >=0.54mmol/L
Advanced glycation end-product，AGEs | Baseline to 4 months
  AGEs are proteins or lipids that become glycated as a result of exposure to sugars. Its can be a factor in aging and in the development from diabetes. The highest value of it means the highest injured did. The data of the post-test should be lower than the data of the pre-test.
Insulin resistance assessment | Baseline to 4 months
  to measure the insulin sensitivity of the cells, the Homeostasis Model Assessment for Insulin Resistance (HOMA-IR) method will be applied in this study. The highest value of it means the highest injured did. The data of the post-test should be lower than the data of the pre-test.
Beta-cell function assessment | Baseline to 4 months
  to measure the function of the Beta-cell, the HOMA-beta-cell method will be applied in this study. The highest value of it means the function of the Beta-cell more normal. The data of the post-test should be higher than the data of the pre-test.
Autonomic nervous system assessment - Heart Rate | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is HR(Heart Rate).
  HR(1/min):normal range(60-100),abnormal range(lower than 60 or higher than 100)
Autonomic nervous system assessment - blood pressure | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about blood pressure.
  SYS(mmHg):normal range(90-140), abnormal range(higher than 140) DIA(mmHg):normal range(60-90), abnormal range(higher than 90) SYS(mmHg) and DIA(mmHg) will be combined to report blood pressure in SYS/DIA(mmHg)
Autonomic nervous system assessment - Heart Rate Variability | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about HRV(Heart Rate Variability).
  HRV(ms): normal range(25-100), abnormal range(lower than 15)
Autonomic nervous system assessment - Low Frequency | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about LF(Low Frequency %).
  LF(%): normal range(40-70), abnormal range(higher than 80)
Autonomic nervous system assessment - High Frequency | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about HF(High Frequency %).
  HF(%): normal range(25-40), abnormal range(lower than 20)
Autonomic nervous system assessment - Low/High Frequency standard | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about LF/HF(Low/High Frequency standard).
  LF/HF: normal range(0.5-2.5), abnormal range(higher than 3)
Autonomic nervous system assessment - Irregular Heartbeat standard | Baseline to 4 months
  the measurement of Autonomic nervous system assessment is to measure the functions of sympathetic and the parasympathetic. The scale of this assessment is about IR(Irregular Heartbeat standard).
  IR: normal range(0-3), abnormal range(higher than 4)
Pittsburgh sleep quality index (PSQI) | Baseline to 4 months
  The PSQI is a questionnaire to measure sleep quality over the past month. the 19 items question can be grouped into 7 components, its (1)sleep duration; (2) sleep disturbance;(3) sleep latency; (4) daytime dysfunction due to sleepiness; (5) sleep efficiency; (6) overall sleep quality; (7) sleep medication use. The sleep component scores are summed to a total score ranging from 0 to 21. The higher of the total score means the sleep quality worse.
Knee Pain - Numeric Rating Scale, Knee Pain - NRS | Baseline to 4 months
  To measure the Knee's painfulness. The higher of the score means the knee's more painful.
Geriatric Depression Scale-15, GDS-15 | Baseline to 4 months
  to assess depressive symptoms among old people with differing level of cognitive function.
  1-5 : healthy 6-9 : light depression 10 and above : serious depression

CONTACTS AND LOCATIONS:
Overall Officials: Ching Yong Chin, Master, Principal Investigator — Nanhua University; Yi-Wen Huang, Master, Principal Investigator — Nanhua University; Jin-Bang Shang, Master, Principal Investigator — Nanhua University
Locations (1):
- Department of Natural Biotechnology, Master's program in Natural Healing Sciences Nanhua University, Dalin, Chiayi, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cegrell L. The occurrence of biogenic monoamines in the mammalian endocrine pancreas. Acta Physiol Scand Suppl. 1968;314:1-60. No abstract available. PMID 4973243
- [Background] Chang Y, Liu YP, Liu CF. The effect on serotonin and MDA levels in depressed patients with insomnia when far-infrared rays are applied to acupoints. Am J Chin Med. 2009;37(5):837-42. doi: 10.1142/S0192415X09007272. PMID 19885944
- [Background] COUPLAND RE. The innervation of pan creas of the rat, cat and rabbit as revealed by the cholinesterase technique. J Anat. 1958 Jan;92(1):143-9. No abstract available. PMID 13513506
- [Background] Dandona P, Aljada A, Bandyopadhyay A. Inflammation: the link between insulin resistance, obesity and diabetes. Trends Immunol. 2004 Jan;25(1):4-7. doi: 10.1016/j.it.2003.10.013. PMID 14698276
- [Background] Giacco F, Brownlee M. Oxidative stress and diabetic complications. Circ Res. 2010 Oct 29;107(9):1058-70. doi: 10.1161/CIRCRESAHA.110.223545. PMID 21030723
- [Background] Haag M, Dippenaar NG. Dietary fats, fatty acids and insulin resistance: short review of a multifaceted connection. Med Sci Monit. 2005 Dec;11(12):RA359-67. Epub 2005 Nov 24. PMID 16319806
- [Background] Haffner SM, Kennedy E, Gonzalez C, Stern MP, Miettinen H. A prospective analysis of the HOMA model. The Mexico City Diabetes Study. Diabetes Care. 1996 Oct;19(10):1138-41. doi: 10.2337/diacare.19.10.1138. PMID 8886564
- [Background] Honda K, Inoue S. Sleep-enhancing effects of far-infrared radiation in rats. Int J Biometeorol. 1988 Jun;32(2):92-4. doi: 10.1007/BF01044900. No abstract available. PMID 3410585
- [Background] Benzie IF, Strain JJ. The ferric reducing ability of plasma (FRAP) as a measure of "antioxidant power": the FRAP assay. Anal Biochem. 1996 Jul 15;239(1):70-6. doi: 10.1006/abio.1996.0292. PMID 8660627
- [Background] Lu FJ, Lin JT, Wang HP, Huang WC. A simple, sensitive, non-stimulated photon counting system for detection of superoxide anion in whole blood. Experientia. 1996 Feb 15;52(2):141-4. doi: 10.1007/BF01923359. PMID 8608815
- [Background] Ishibashi J, Yamashita K, Ishikawa T, Hosokawa H, Sumida K, Nagayama M, Kitamura S. The effects inhibiting the proliferation of cancer cells by far-infrared radiation (FIR) are controlled by the basal expression level of heat shock protein (HSP) 70A. Med Oncol. 2008;25(2):229-37. doi: 10.1007/s12032-007-9020-4. Epub 2007 Oct 30. PMID 17968683
- [Background] Kahn SE, Hull RL, Utzschneider KM. Mechanisms linking obesity to insulin resistance and type 2 diabetes. Nature. 2006 Dec 14;444(7121):840-6. doi: 10.1038/nature05482. PMID 17167471
- [Background] Kasznicki J, Kosmalski M, Sliwinska A, Mrowicka M, Stanczyk M, Majsterek I, Drzewoski J. Evaluation of oxidative stress markers in pathogenesis of diabetic neuropathy. Mol Biol Rep. 2012 Sep;39(9):8669-78. doi: 10.1007/s11033-012-1722-9. Epub 2012 Jun 21. PMID 22718504
- [Background] Lin CC, Chiang YS, Lung CC. Effect of infrared-C radiation on skin temperature, electrodermal conductance and pain in hemiparetic stroke patients. Int J Radiat Biol. 2015 Jan;91(1):42-53. doi: 10.3109/09553002.2014.937512. Epub 2014 Aug 11. PMID 24991883
- [Background] Maritim AC, Sanders RA, Watkins JB 3rd. Diabetes, oxidative stress, and antioxidants: a review. J Biochem Mol Toxicol. 2003;17(1):24-38. doi: 10.1002/jbt.10058. PMID 12616644
- [Background] Masuda A, Kihara T, Fukudome T, Shinsato T, Minagoe S, Tei C. The effects of repeated thermal therapy for two patients with chronic fatigue syndrome. J Psychosom Res. 2005 Apr;58(4):383-7. doi: 10.1016/j.jpsychores.2004.11.005. PMID 15992574
- [Background] Matthews DR, Hosker JP, Rudenski AS, Naylor BA, Treacher DF, Turner RC. Homeostasis model assessment: insulin resistance and beta-cell function from fasting plasma glucose and insulin concentrations in man. Diabetologia. 1985 Jul;28(7):412-9. doi: 10.1007/BF00280883. PMID 3899825
- [Background] Riccardi G, Giacco R, Rivellese AA. Dietary fat, insulin sensitivity and the metabolic syndrome. Clin Nutr. 2004 Aug;23(4):447-56. doi: 10.1016/j.clnu.2004.02.006. PMID 15297079
- [Background] Saito M, Marumo K. Effects of Collagen Crosslinking on Bone Material Properties in Health and Disease. Calcif Tissue Int. 2015 Sep;97(3):242-61. doi: 10.1007/s00223-015-9985-5. Epub 2015 Mar 20. PMID 25791570
- [Background] Saslow L, Mason AE, Kim S, Goldman V, Ploutz-Snyder R, Bayandorian H, Daubenmier J, Hecht FM, Moskowitz JT. Authors' Reply: Comment on "An Online Intervention Comparing a Very Low-Carbohydrate Ketogenic Diet and Lifestyle Recommendations Versus a Plate Method Diet in Overweight Individuals With Type 2 Diabetes: A Randomized Controlled Trial". J Med Internet Res. 2018 May 1;20(5):e181. doi: 10.2196/jmir.8776. No abstract available. PMID 29716886
- [Background] Stratton IM, Adler AI, Neil HA, Matthews DR, Manley SE, Cull CA, Hadden D, Turner RC, Holman RR. Association of glycaemia with macrovascular and microvascular complications of type 2 diabetes (UKPDS 35): prospective observational study. BMJ. 2000 Aug 12;321(7258):405-12. doi: 10.1136/bmj.321.7258.405. PMID 10938048
- [Background] Tahrani AA, Piya MK, Kennedy A, Barnett AH. Glycaemic control in type 2 diabetes: targets and new therapies. Pharmacol Ther. 2010 Feb;125(2):328-61. doi: 10.1016/j.pharmthera.2009.11.001. Epub 2009 Nov 18. PMID 19931305
- [Background] Toyokawa H, Matsui Y, Uhara J, Tsuchiya H, Teshima S, Nakanishi H, Kwon AH, Azuma Y, Nagaoka T, Ogawa T, Kamiyama Y. Promotive effects of far-infrared ray on full-thickness skin wound healing in rats. Exp Biol Med (Maywood). 2003 Jun;228(6):724-9. doi: 10.1177/153537020322800612. PMID 12773705
- [Background] Yu SY, Chiu JH, Yang SD, Hsu YC, Lui WY, Wu CW. Biological effect of far-infrared therapy on increasing skin microcirculation in rats. Photodermatol Photoimmunol Photomed. 2006 Apr;22(2):78-86. doi: 10.1111/j.1600-0781.2006.00208.x. PMID 16606412
- [Result] Beever R. Far-infrared saunas for treatment of cardiovascular risk factors: summary of published evidence. Can Fam Physician. 2009 Jul;55(7):691-6. PMID 19602651
- [Result] Burleson MH, Malarkey WB, Cacioppo JT, Poehlmann KM, Kiecolt-Glaser JK, Berntson GG, Glaser R. Postmenopausal hormone replacement: effects on autonomic, neuroendocrine, and immune reactivity to brief psychological stressors. Psychosom Med. 1998 Jan-Feb;60(1):17-25. doi: 10.1097/00006842-199801000-00004. PMID 9492234